CLINICAL TRIAL: NCT02976558
Title: Prospective Open Randomized Monocentric Two-armed Controlled Clinical Trial in Parallel Groups to Investigate the Influence of Complementary Medicine (CAM) Interventions on Quality of Life and The Treatment Process of Patients Undergoing Allogenic Stem Cell Transplantation
Brief Title: The Influence of TaKeTiNa Music Therapy, Traditional Chinese Acupuncture and Clown Theatrical Performance on Quality of Life and the Therapeutic Process of Patients Undergoing Allogenic Stem Cell Transplantation
Acronym: TriCAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to organisational issues, the study had to be completed prematurely.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ali Behzad, Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCS Erlangen 0383
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Hematological Neoplasm; Graft-Versus-Host Disease; Depression; Stem Cell Transplant Complications; Quality of Life; Leukemia
Keywords: CAM; allogenic Stem Cell Transplantation; Graft-Versus-Host Disease; Depression; Quality of Life; Acupuncture; Traditional chinese Medicine; Integrative medicine; Complementary and Alternative Medicine; Music therapy TaKeTiNa; Clown theatrical performance; Humour; Chemotherapy side effects; Psycho neuro immune system; GvHD; PNEIS; CMV; EBV; holistic medicine
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease; Depression; Leukemia | interventions — Health; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Interventions:
  Acupuncture, music therapy (TaKeTiNa) and Clown theatrical performance starting before allogenic stem cell transplant until three months after transplantation.
  Interventions each twice a week for 4 weeks, then once a week for 4 weeks, then once every two weeks for 4 weeks
  Interventions: Behavioral: Clown theatrical Performance; Procedure: Acupuncture; Behavioral: Music Therapy TaKeTiNa
- Control Group (No Intervention): control group. No interventions

INTERVENTIONS:
Behavioral: Clown theatrical Performance
  Other Names: theatre therapy, humour for health
  Arms: Treatment Group
Procedure: Acupuncture — Acupuncture according to Traditional Chinese Medicine
  Arms: Treatment Group
Behavioral: Music Therapy TaKeTiNa
  Arms: Treatment Group

SUMMARY:
The allogenic stem cell transplantation (aSCT), the only curative approach for many hematological diseases, often leads to severe diseases or chronic conditions, leaving patients with physical disabilities and severe depression and impacting their quality of life in many cases. These consequences are still not adequately addressed by conventional therapies. In this study, the investigators examine the influence of the three complementary medicine methods (CAM) namely acupuncture according to Traditional Chinese Medicine (TCM), music therapy according to the TaKeTiNa method and the psychological disease processing by theatrical clown performance on the quality of life and the therapy process of patients before and after aSCT.

DETAILED DESCRIPTION:
The allogenic stem cell transplantation (aSCT) is still the only curative approach for many hematological diseases. Despite new therapeutic developments in the past few years, the therapy-associated mortality rate is around 20%. Patients develop a Graft versus Host Disease (GvHD) in 30-70% of the cases, some with persistent, severe progression and often complicated by infections. In severe chronic conditions, physical disabilities such as weakness, paralysis, scarred vulnerable skin, and blindness may occur. A significant reduction in the quality of life of these patients including severe depression is the consequence.

The demand of patients for supplementary therapy possibilities in the sense of an integrative, complementary medicine is great. There are indications that complementary methods can help improve the quality of life and reduce the associated side effects. However, there are no scientific studies to clarify the efficacy or safety of such therapies in the aSCT.

In this project, the investigators examine the influence of three complementary medicine methods, namely acupuncture according to Traditional Chinese Medicine (TCM), music therapy according to the TaKeTiNa method and the psychological disease processing by theatrical clown performance, on the quality of life and the therapy process of patients before and after aSCT.

Acupuncture according to TCM is an evidence-based therapy approach with few side effects for many diseases. In the past few years, not only their superiority over placebo treatment, but also the point-specific effect has been shown. Based on the numerous published data on pain, nausea, fatigue and depression, it can be assumed that acupuncture reduces the side effects of drug therapy in aSCT and thus improves the quality of life of patients.

According to TCM, the points influence the flow of the energy (referred to as "Qi") in the body and stimulate its self-regulation. In addition, each organ system associated to a different emotion. The unimpeded flow of the ongoing arising of emotions and body energies is, according to TCM, a prerequisite for the health of the organism.

In TCM, the acupuncture used to stimulate the self-regulation of the body is accompanied by the regular practice of Qi-Gong or Tai-Qi by the patient to achieve the greatest therapeutic effect between the treatments. This additive component can hardly be realized because of the severely restricted general state of the patients.

In order to mobilize the energy and emotions, this study also implements two further treatment modalities, which are practiced with the patient and which the patient can practice on a daily basis by himself:

TaKeTiNa is a form of music therapy founded by Reinhard Flatischler, in which body, voice and movement are used to develop present consciousness, physical feeling and rhythm skills. It has been used therapeutically for more than 20 years.

Furthermore, the processing of arising emotions needs to be facilitated. Patients undergoing an aSCT are exposed to a deeply invasive and debilitating situation for a period of at least four weeks. Characteristics are social isolation through limited visits as well as confinement to a small room, almost complete loss of the privacy and independence through frequent monitoring and lavation necessary during aSCT. Finally the confrontation with the illness, the side effects of the drug treatment and the possible death. Arising emotions can lead to a blockade in the energy flow of the respective organ according to TCM and can cause illness. Therefore, the introduction of six basic gestures from the clown performance according to the Metzler method (KANA-Institut für Koerperprache Freiburg) is intended to give the patient the opportunity to process his emotions in a playful manner in real time or to communicate them directly to another person without words.

ELIGIBILITY:
Inclusion Criteria:

* planned allogenic stem cell transplantation
* patient mentally and intellectually able to understand and sign the form

Exclusion Criteria:

* Current enrollment in another intervention study
* clinical diagnosis of depression by HADS-D score plus drug therapy for depression at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Difference in the Quality of Life of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through FACT-G Questionaire

SECONDARY OUTCOMES:
Difference in development of GvHD of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through staging of GvHD and required days of hospitalisation
Difference in development of fungal infections of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through required days of hospitalisation and antimycotic therapy
Difference in development of bacterial infections of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through required days of hospitalisation and antibiotic therapy
Difference in development of viral infections including CMV and EBV of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through required days of hospitalisation and antiviral therapy
Difference in Depression of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through HADS-D questionaire
Impact of the diagnosis and therapy according to traditional chinese medicine on the difference in development of Infections of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment days of hospitalisation and antiinfective therapy
Impact of the diagnosis and therapy according to traditional chinese medicine on the difference in development of GvHD of the intervention group compared to the control group | day 1 of study compared to day 90 of study
  Assessment through staging of GvHD and required days of hospitalisation
Impact on the development of hematoma and soft tissue infections that need treatment (2nd Amendment) | from day 1 of study to day 90
  Patients in the intervention group receive acupuncture as one of the three treatment modalities. Any development of hematoma on the skin or any soft tissue infection that need either local treatment (cooling agents, medical ointments etc.) or systemic treatment (surgery or systemic antibiotics) will be documented as an event. Total number of hematomas needing treatment and soft tissue infections needing treatment will be compared between intervention and control group

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen Nuermberg Medical School, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Bacigalupo A, Sormani MP, Lamparelli T, Gualandi F, Occhini D, Bregante S, Raiola AM, di Grazia C, Dominietto A, Tedone E, Piaggio G, Podesta M, Bruno B, Oneto R, Lombardi A, Frassoni F, Rolla D, Rollandi G, Viscoli C, Ferro C, Garbarino L, Van Lint MT. Reducing transplant-related mortality after allogeneic hematopoietic stem cell transplantation. Haematologica. 2004 Oct;89(10):1238-47. PMID 15477210
- [Background] Blazar BR, Murphy WJ, Abedi M. Advances in graft-versus-host disease biology and therapy. Nat Rev Immunol. 2012 May 11;12(6):443-58. doi: 10.1038/nri3212. PMID 22576252
- [Background] Braamse AM, Yi JC, Visser OJ, Heymans MW, van Meijel B, Dekker J, Syrjala KL. Developing a Risk Prediction Model for Long-Term Physical and Psychological Functioning after Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2016 Mar;22(3):549-56. doi: 10.1016/j.bbmt.2015.11.1102. Epub 2015 Dec 11. PMID 26685773
- [Background] Fasching PA, Thiel F, Nicolaisen-Murmann K, Rauh C, Engel J, Lux MP, Beckmann MW, Bani MR. Association of complementary methods with quality of life and life satisfaction in patients with gynecologic and breast malignancies. Support Care Cancer. 2007 Nov;15(11):1277-1284. doi: 10.1007/s00520-007-0231-1. Epub 2007 Mar 1. PMID 17333294
- [Background] Garcia MK, McQuade J, Haddad R, Patel S, Lee R, Yang P, Palmer JL, Cohen L. Systematic review of acupuncture in cancer care: a synthesis of the evidence. J Clin Oncol. 2013 Mar 1;31(7):952-60. doi: 10.1200/JCO.2012.43.5818. Epub 2013 Jan 22. PMID 23341529
- [Background] Lee A, Chan SK, Fan LT. Stimulation of the wrist acupuncture point PC6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2015 Nov 2;2015(11):CD003281. doi: 10.1002/14651858.CD003281.pub4. PMID 26522652
- [Background] Shneerson C, Taskila T, Gale N, Greenfield S, Chen YF. The effect of complementary and alternative medicine on the quality of life of cancer survivors: a systematic review and meta-analyses. Complement Ther Med. 2013 Aug;21(4):417-29. doi: 10.1016/j.ctim.2013.05.003. Epub 2013 Jun 3. PMID 23876573
- [Background] Sun CL, Francisco L, Baker KS, Weisdorf DJ, Forman SJ, Bhatia S. Adverse psychological outcomes in long-term survivors of hematopoietic cell transplantation: a report from the Bone Marrow Transplant Survivor Study (BMTSS). Blood. 2011 Oct 27;118(17):4723-31. doi: 10.1182/blood-2011-04-348730. Epub 2011 Aug 5. PMID 21821714
- [Background] Saramago P, Woods B, Weatherly H, Manca A, Sculpher M, Khan K, Vickers AJ, MacPherson H. Methods for network meta-analysis of continuous outcomes using individual patient data: a case study in acupuncture for chronic pain. BMC Med Res Methodol. 2016 Oct 6;16(1):131. doi: 10.1186/s12874-016-0224-1. PMID 27716074
- [Background] Witt CM, Pach D, Brinkhaus B, Wruck K, Tag B, Mank S, Willich SN. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. Forsch Komplementmed. 2009 Apr;16(2):91-7. doi: 10.1159/000209315. Epub 2009 Apr 9. PMID 19420954
- [Background] Fuentealba Cargill F, Biagini Alarcon L. [Acupuncture for postoperative pain, a literature review]. Rev Med Chil. 2016 Mar;144(3):325-32. doi: 10.4067/S0034-98872016000300007. Spanish. PMID 27299818